CLINICAL TRIAL: NCT05221749
Title: The Antibacterial Effect of Nanosilver Fluoride in Relation to Caries Activity in Primary Teeth: a Randomized Controlled Clinical Trial
Brief Title: The Antibacterial Effect of Nanosilver Fluoride on Primary Teeth
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Only the 1 month follow-up was completed. The principal investigator could not complete the 3 month follow-up appointments and was not calibrated with other dentists who were available at the time.
Sponsor: Nour Ammar, BDS (Other)
Responsible Party: Sponsor-Investigator, Nour Ammar, BDS, Instructor, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AlexandriaU1
Record Dates: First submitted 2021-12-25; First posted 2022-02-03 (Actual); Results first posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-07

CONDITIONS: Primary Teeth; Microbial Colonization; Caries; Dental Caries in Children
Keywords: Nano silver fluoride; silver diamine fluoride; antibacterial; caries arrest; microbiology; primary teeth; pediatric; clinical trial; nanosilver; SDF
MeSH Terms: conditions — Communicable Diseases | interventions — silver diamine fluoride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Silver diamine fluoride (Active Comparator): These active caries lesions will receive silver diamine fluoride treatment
  Interventions: Drug: Silver diamine fluoride
- Nanosilver fluoride (Experimental): These active caries lesions will receive nanosilver fluoride treatment
  Interventions: Drug: Nanosilver Fluoride (NSF)

INTERVENTIONS:
Drug: Nanosilver Fluoride (NSF) — Optimized synthesis of Nanosilver Fluoride
  Other Names: Nanosilver Fluoride
  Arms: Nanosilver fluoride
Drug: Silver diamine fluoride — Silver Diamine Fluoride
  Other Names: Advantage Arrest by Elevate Oral care, 38% SDF
  Arms: Silver diamine fluoride

SUMMARY:
To assess the antibacterial effect of Nanosilver Fluoride (NSF) in relation to caries activity in dentin caries lesions of primary teeth in comparison to Silver Diamine Fluoride (SDF).

DETAILED DESCRIPTION:
Fifty children aged 4 to 6 years old with active dentin caries lesions (score 5 according to International Detection and Assessment System (ICDAS II) criteria) will be enrolled in the study. They will be equally and randomly allocated into 2 groups: a group receiving NSF and a control group receiving SDF treatment. Microbiological samples will be collected from the carious lesions and from unstimulated saliva at the baseline and at the 1 and 3 months' follow-up appointments. Bacterial counts will be assessed using Mitis Salivarius agar (selective culture media for S. mutans) and Rogosa agar (selective culture media for lactobacilli), and the results will be expressed in colony-forming units. Data regarding the children's oral health will be collected and their dmf index will be scored. The arrest of active carious lesions will be measured at the follow-up appointments according to ICDAS II criteria.

ELIGIBILITY:
Inclusion Criteria:

* The presence of at least one active carious lesion on a primary tooth.
* Completion of an informed consent to participate in the study.

Exclusion criteria:

* Children reporting spontaneous or elicited pain from caries or showing any signs of pulpal infection, swelling, abscess, obvious discoloration of the tooth, or premature mobility.
* Reported usage of local or systemic antibiotics, chlorhexidine or fluoride mouthwashes within the last 2 weeks.
* Children presenting with special health care needs or undergoing medical treatment for chronic or acute diseases affecting salivary flow.
* Allergy or sensitivity to silver or any of the materials included in the study.
* Child weight less than 10 Kg (to avoid concerns for toxicity).

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nour Ammar, BDS, Principal Investigator — Faculty of dentistry, Alexandria University, Alexandria, Egypt.
Locations (1):
- Faculty of Dentistry, Alexandria Univeristy, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
Each participant will be provided with a serial number that will only be accessible to the principal investigator. No data regarding the identity of the participants will be shared under any circumstances. All participants or their guardians must provide a written informed consent prior to any procedures.

REFERENCES:
- [Derived] Ammar N, El-Tekeya MM, Talat DM, Essa S, Essawy MM, Kuhnisch J, Hamed H, Nabil N, Achy SE, Tantawi ME. Effect of silver diamine fluoride and nanosilver on salivary bacterial counts in children with early childhood caries: a randomized controlled clinical trial. BMC Oral Health. 2025 Jun 9;25(1):945. doi: 10.1186/s12903-025-06325-3. PMID 40490725
- [Derived] Ammar N, El-Tekeya MM, Essa S, Essawy MM, Talaat DM. Antibacterial effect and impact on caries activity of nanosilver fluoride and silver diamine fluoride in dentin caries of primary teeth: a randomized controlled clinical trial. BMC Oral Health. 2022 Dec 30;22(1):657. doi: 10.1186/s12903-022-02697-y. PMID 36585664
- [Derived] Ammar N, El-Tekeya MM, Essa S, Essawy MM, El Achy SN, Talaat DM. The antibacterial effect of nanosilver fluoride in relation to caries activity in primary teeth: a protocol for a randomized controlled clinical trial. Trials. 2022 Jul 8;23(1):558. doi: 10.1186/s13063-022-06477-5. PMID 35804457

RESULTS

PARTICIPANT FLOW:
Groups:
- Silver Diamine Fluoride (SDF): These active caries lesions will receive one application of 38% silver diamine fluoride at the baseline appointment.
- Nanosilver Fluoride (NSF): These active caries lesions will receive one application of nanosilver fluoride at the baseline appointment.
Period: Overall Study
Arm/Group | Silver Diamine Fluoride (SDF) | Nanosilver Fluoride (NSF)
Started | 25 | 25
Completed | 23 | 22
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Population: Children 4-6 years old with at least 1 active dentin caries lesion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Silver Diamine Fluoride | Nanosilver Fluoride | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 25 | 50
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.6 (0.6) | 4.9 (0.9) | 4.75 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 14 | 12 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Egypt | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Antibacterial Effect in Active Dental Caries Lesions
Description: Measuring the percent change in prevalence of cariogenic bacteria using standard microbiological culturing methods, outcome assessment will be done using colony forming units (CFU) from every sample collected. Samples will be collected immediately before application of the intervention (baseline) and one month after the intervention application (1 month follow-up).
  The CFU counts will be used to calculate the percentage change in bacterial prevalence which will be used for assessment and reporting results
Time Frame: 1 month
Measure: Median (Inter-Quartile Range); unit: CFU/mL
Groups:
- Silver Diamine Fluoride (SDF): These active caries lesions will receive silver diamine fluoride treatment
- Nanosilver Fluoride (NSF): These active caries lesions will receive nanosilver fluoride treatment
Arm/Group | Silver Diamine Fluoride (SDF) | Nanosilver Fluoride (NSF)
Number analyzed (Participants) | 25 | 25
CFU/mL
  Baseline | 70000 [1 to 7] | 50000 [1 to 8]
  Follow-up | 20000 [1 to 2] | 5000 [1 to 2]

2. Primary Outcome: The Relation Between the Antibacterial Activity and the Caries Activity in Dental Caries Lesions
Description: A statistical analysis will be done to correlate between the change in number of available cariogenic bacteria from baseline to 1 month (measured in colony forming units) and the caries activity of the lesion (as specified by the international caries detection and assessment system (ICDAS II) criteria.
Time Frame: 1 month
Population: This investigation and consequent analysis were not conducted.
Arm/Group | Silver Diamine Fluoride (SDF) | Nanosilver Fluoride (NSF)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Antibacterial Effect in Unstimulated Saliva Samples
Description: Measuring the change in prevalence of cariogenic bacteria using standard microbiological culturing methods, outcome assessment will be done using colony forming units (CFU) from every sample collected. Samples will be collected before and after the intervention application.
Time Frame: 1 months
Population: This investigation and consequent analysis were not conducted.
Arm/Group | Silver Diamine Fluoride (SDF) | Nanosilver Fluoride (NSF)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: The Relation Between the Antibacterial Activity and the Caries Activity in Dental Caries Lesions
Description: A statistical analysis will be done to correlate between the change in number of available cariogenic bacteria from baseline to 3 months (measured in colony forming units) and the caries activity of the lesion (as specified by the international caries detection and assessment system (ICDAS II) criteria.
Time Frame: 3 month
Population: This investigation and consequent analysis were not conducted.
Arm/Group | Silver Diamine Fluoride (SDF) | Nanosilver Fluoride (NSF)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Antibacterial Effect in Active Dental Caries Lesions
Description: Measuring the change in prevalence of cariogenic bacteria from baseline to 3 months using standard microbiological culturing methods, outcome assessment will be done using colony forming units (CFU) from every sample collected. Samples will be collected before and after the intervention application.
Time Frame: 3 month
Population: This investigation and consequent analysis were not conducted.
Arm/Group | Silver Diamine Fluoride (SDF) | Nanosilver Fluoride (NSF)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Antibacterial Effect in Unstimulated Saliva Samples
Description: as for outcome 5
Time Frame: 3 months
Population: This investigation and consequent analysis were not conducted.
Arm/Group | Silver Diamine Fluoride (SDF) | Nanosilver Fluoride (NSF)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: Participant's carers were contacted within a day of the baseline appointment where the intervention was applied to ask about any side effects or unusual occurrences that may have occurred. However, no side effects were reported for both agents.
Arm/Group | Silver Diamine Fluoride (SDF) | Nanosilver Fluoride (NSF)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT05221749/Prot_SAP_001.pdf